CLINICAL TRIAL: NCT06773156
Title: Sequential Adebrelimab Combined With Apatinib as Consolidation Therapy Following Concurrent Chemoradiotherapy in Limited-Stage Small Cell Lung Cancer: A Prospective, Single-Arm, Multicenter Phase II Clinical Study
Brief Title: Adjuvant Adebrelimab Plus Apatinib After Chemoradiation in Limited-Stage Small Cell Lung Cancer
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Long Huang, Associate Chief Physician of Oncology Department, Second Affiliated Hospital of Nanchang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-SCLC-Ⅱ-021
Record Dates: First submitted 2025-01-03; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Limited-stage Small Cell Lung Cancer (LS-SCLC)
Keywords: Small Cell Lung Cancer; Adebrelimab; Apatinib; Chemoradiation
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adjuvant Adebrelimab Plus Apatinib After Chemoradiation (Experimental)
  Interventions: Drug: Adebrelimab + Apatinib

INTERVENTIONS:
Drug: Adebrelimab + Apatinib — Adebrelimab: Administered by intravenous infusion at a fixed dose of 1200 mg. The infusion should be completed within 30-60 minutes, with a maximum duration of 2 hours. The first dose is given on Day 1, with subsequent doses repeated every 3 weeks. Dose adjustments (either up or down) are not allowed during the study. A maximum delay of 9 weeks for treatment is allowed, or treatment may be terminated.
  Apatinib: 250 mg, taken orally after meals, once daily, continuously. The investigator may temporarily pause the dose or adjust the administration schedule based on symptomatic treatment, such as changing to an every-other-day (qod) schedule or a 5-day-on, 2-day-off regimen. Once toxicity resolves, treatment may resume at the original dose.
  The combined treatment of Adebrelimab + Apatinib for consolidation therapy should not exceed 24 months in total.

SUMMARY:
The study includes the screening period (from the time the subject signs the informed consent form to no more than 28 days before the first dose, imaging evaluations are allowed within 28 days before the first dose, and 5-14 days after the last radiotherapy/chemotherapy treatment, as close as possible to the treatment start date and the start of the study treatment), tumor tissue biopsy collection based on the subject's hospital, with preferred samples obtained within ≤3 months, but archived samples within 6 months before the first dose are also acceptable. The treatment period (until disease progression/worsening or confirmed radiological disease progression, or withdrawal for any reason) and the follow-up period (from the last dose to 36 months, including safety follow-up and survival follow-up).

**Screening Period:** Subjects who have received 2-4 cycles of platinum-based concurrent or induction chemotherapy (cCRT) and are evaluated as having non-progressive disease after cCRT, with the cCRT treatment ending within 1-42 days before the first dose, and the last radiotherapy session as the final end time. Consolidation chemotherapy after radiotherapy is not allowed.

Screening evaluation must be performed within 28 days before the first dose to determine eligibility. Tumor tissue samples should be collected based on the subject's hospital. The preferred samples are archived or freshly obtained tumor tissue wax blocks or pathological biopsy slides within ≤3 months, but archived samples within 6 months before the first dose are also acceptable.

**Treatment Period:** Each treatment cycle is 3 weeks. Atezolizumab 1200mg is administered via intravenous infusion, and Apatinib 250mg is taken orally after meals, once daily, for continuous use.

Subjects must undergo a comprehensive examination at the end of the study treatment or when withdrawing from the study, including vital signs, physical examination, laboratory tests, quality of life assessment, clinical tumor imaging evaluation (CT or MRI), and other necessary checks.

**Follow-up Period:** After the study treatment ends or the subject withdraws from the study, safety follow-up should be conducted. Subjects should be followed up every 30±7 days until 90 days. The first (30±7 days after withdrawal from the group) safety visit must be conducted at the research center, and vital signs, physical examination, laboratory tests, etc., should be assessed for AEs, concomitant medications, and supportive treatments. The other two visits (60±7 days and 90±7 days after withdrawal from the group) will be conducted by telephone, collecting survival information, AEs, concomitant medications, and supportive treatments.

After the safety follow-up is completed, subjects will be followed up every 3 months by phone to monitor survival status until death, loss to follow-up, withdrawal of informed consent, observation for 3 years, or termination of the study.

DETAILED DESCRIPTION:
Dosing Regimen： Adebrelimab:Administered by intravenous infusion at a fixed dose of 1200 mg. The infusion should be completed within 30-60 minutes, with a maximum duration of 2 hours. The first dose is given on Day 1, with subsequent doses repeated every 3 weeks. Dose adjustments (either up or down) are not allowed during the study. A maximum delay of 9 weeks for treatment is allowed, or treatment may be terminated.

Apatinib: 250 mg, taken orally after meals, once daily, continuously. The investigator may temporarily pause the dose or adjust the administration schedule based on symptomatic treatment, such as changing to an every-other-day (qod) schedule or a 5-day-on, 2-day-off regimen. Once toxicity resolves, treatment may resume at the original dose.

The combined treatment of Adebrelimab + Apatinib for consolidation therapy should not exceed 24 months in total.

Primary Outcome Measure Progression-free survival (PFS) as assessed by the investigator (according to RECIST 1.1).

Secondary Outcome Measures

1. Efficacy:Overall survival (OS), 12-month/24-month/36-month OS rates, 12-month/18-month PFS rates (according to RECIST 1.1).
2. Safety: Including treatment-related adverse events (AEs), serious adverse events (SAEs), and the incidence of AEs and SAEs related to the study drugs (assessed based on the NCI CTCAE 5.0 criteria).
3. Quality of Life (QoL): Changes in symptoms, functions, and overall health status/QoL reported by the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years (inclusive), gender unrestricted;
* Histologically confirmed limited-stage small cell lung cancer (SCLC), not previously treated with systemic antitumor therapy (defined as stage I-III according to the American Joint Committee on Cancer 8th edition, with all lesions manageable within a tolerable radiation therapy plan);
* ECOG performance status (PS) of 0 or 1;
* Received radical concurrent or induction chemoradiotherapy, achieving complete response (CR), partial response (PR), or stable disease (SD) after cCRT. The chemotherapy regimen includes platinum-based drugs and etoposide, with 2-4 cycles of chemotherapy. Radiation therapy doses are 60-66 Gy QD (2 Gy per fraction) or 45 Gy BID (1.5 Gy per fraction). No disease progression after chemoradiation; whether prophylactic cranial irradiation (PCI) is performed will be decided by the investigator, and PCI should be completed within 1-42 days after chemoradiation. The first dose of the study drug should be administered within 1-42 days after chemoradiation;
* Based on the subject's consent, blood samples should be provided or collected for biomarker analysis after concurrent chemoradiation and consolidation therapy;
* Laboratory test results meet the following conditions, with adequate hematologic and organ function: a) Complete blood count: Absolute neutrophil count (ANC) ≥1.5 × 10^9/L, with no use of granulocyte colony-stimulating factor support within 14 days prior to the first dose; lymphocyte count (LC) ≥0.5 × 10^9/L; platelet count (PLT) ≥100 × 10^9/L; hemoglobin (Hb) ≥90 g/L, with no blood transfusion within 14 days prior to the first dose; b) Liver function: Aspartate transaminase (AST) and alanine transaminase (ALT) ≤3 × ULN; total bilirubin (TBIL) ≤1.5 × ULN (for patients with diagnosed Gilbert's syndrome, total bilirubin ≤3.0 mg/dL); alkaline phosphatase (ALP) ≤2.5 × ULN; albumin (ALB) ≥3 g/dL; c) Renal function: Creatinine clearance rate (CrCl) ≥45 mL/min (for carboplatin group); CrCl ≥60 mL/min (for cisplatin group) (CrCl can be calculated using the Cockcroft-Gault formula, Chronic Kidney Disease Epidemiology Collaboration formula, or Modification of Diet in Renal Disease formula). Urinary protein <2+ (if urinary protein ≥2+, a 24-hour urinary protein quantification test should be performed, and subjects with 24-hour urinary protein <1g are eligible for the study); d) Coagulation function: International normalized ratio (INR) ≤1.5, activated partial thromboplastin time (APTT) ≤1.5 × ULN;
* Pulmonary function tests: Forced expiratory volume in 1 second (FEV1) >50% of predicted normal value, and diffusion capacity of the lungs for carbon monoxide (DLCO) or transfer factor of the lungs for carbon monoxide (TLCO) >40% of predicted normal value; if the subject does not meet these criteria but has clinical indications, treatment with inhaled corticosteroids and bronchodilators may be administered, and reevaluation should be performed 1-2 weeks later to determine eligibility;
* Non-surgically sterilized females of childbearing potential or male subjects must agree to use at least one medically approved contraceptive method (such as intrauterine device or oral contraceptives) during the study and for 3 months after the study treatment period; non-surgically sterilized females of childbearing potential must have a negative serum HCG test within 7 days prior to the first dose;
* Non-surgically sterilized females of childbearing potential or male subjects must agree to use at least one medically approved contraceptive method (such as intrauterine device or oral contraceptives) during the study and for 3 months after the study treatment period; non-surgically sterilized females of childbearing potential must have a negative serum HCG test within 7 days prior to the first dose.

Exclusion Criteria:

* Histopathologically confirmed mixed-type SCLC or NSCLC (mixed component > 10%);
* Previous systemic anti-tumor therapy for SCLC or treatment with immune checkpoint inhibitors, as well as any systemic therapy targeting VEGF or VEGFR; if the patient has previously received traditional Chinese medicine (TCM) for anti-tumor treatment, there must be at least a 2-week interval between the end of TCM treatment and the first dose of the study drug;
* Extensive-stage SCLC;
* Operable SCLC (clinical stage T1-2N0, except for those with surgical contraindications or who refuse surgery);
* Participation in another clinical study within 28 days prior to the first dose of the investigational drug, or use of any investigational drug;
* Presence of malignant pleural effusion. If the patient has drainable pleural effusion during screening, at least one thoracentesis must be performed to confirm the presence of malignant cells;
* Known or suspected interstitial lung disease; other moderate to severe pulmonary diseases that may interfere with the detection or management of drug-related pulmonary toxicity, including but not limited to idiopathic pulmonary fibrosis, organizing pneumonia/bronchiolitis obliterans, etc.;
* Active, known, or suspected autoimmune diseases or a history of autoimmune diseases, including but not limited to myasthenia gravis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, etc. Patients with type I diabetes (well-controlled with insulin therapy), residual hypothyroidism due to autoimmune thyroiditis requiring only hormone replacement therapy, or conditions not expected to recur in the absence of external triggers may be enrolled. Patients with eczema, psoriasis, chronic lichen simplex, or vitiligo (excluding psoriatic arthritis) with skin rash covering less than 10% of the body surface area, well-controlled at baseline, and requiring only low-potency topical steroids, without acute exacerbation of the underlying condition in the past 12 months (no PUVA, methotrexate, retinoids, biologics, oral calcineurin inhibitors, high-potency or oral steroids), may be included;
* Concurrent malignancies within ≤5 years prior to the first dose, except for adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, localized prostate cancer after radical surgery, or ductal carcinoma in situ after radical surgery (hormonal therapy for non-metastatic prostate or breast cancer is allowed);
* Significant clinical history of cardiovascular or cerebrovascular diseases, including but not limited to: (1) congestive heart failure (NYHA class ≥2); (2) unstable angina or clinically significant ventricular arrhythmia requiring intervention within 1 month prior to the first dose; (3) myocardial infarction or cerebrovascular accident within 3 months prior to signing the ICF; (4) left ventricular ejection fraction (LVEF) <50% within 28 days prior to the first dose;
* Arterial/venous thrombotic events within 6 months prior to the first dose, such as deep vein thrombosis or pulmonary embolism;
* Hypertension that cannot be adequately controlled with antihypertensive therapy (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg);
* Clinically significant bleeding symptoms or clear evidence of bleeding tendency within 3 months prior to the first dose, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood ≥++, or vasculitis, regardless of severity;
* Significant hemoptysis or daily hemoptysis ≥2.5 mL within 30 days prior to the first dose;
* Known hereditary or acquired bleeding or thrombotic tendencies (e.g., hemophilia, coagulation disorders, thrombocytopenia, hypersplenism, etc.);
* Urinalysis showing proteinuria ≥(++) or 24-hour urinary protein ≥1.0 g;
* Severe infections within 4 weeks prior to the first dose, including but not limited to bacteremia or severe pneumonia requiring hospitalization; active infections requiring systemic antibiotic therapy with CTCAE ≥2 within 2 weeks prior to the first dose;
* Evidence of active tuberculosis infection within 1 year prior to the first dose, or a history of active tuberculosis more than 1 year ago without standard treatment;
* History of immunodeficiency, including positive HIV serology;
* Active hepatitis B [defined as positive hepatitis B surface antigen (HBsAg) at screening with HBV-DNA levels above the upper limit of normal (ULN) at the local laboratory (if no ULN is available, HBV-DNA must be <1000 copies/mL or 500 IU/mL)] or hepatitis C [defined as positive hepatitis C antibody (HCV-Ab) at screening with positive HCV-RNA];
* Systemic immunosuppressive therapy within 14 days prior to the first dose (including but not limited to glucocorticoids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF drugs); patients receiving short-term, systemic immunosuppressive therapy (e.g., glucocorticoids for nausea, vomiting, or allergic reactions) may be discussed with the investigator for eligibility. Inhaled glucocorticoids for chronic obstructive pulmonary disease, mineralocorticoids (e.g., fludrocortisone) for orthostatic hypotension, and low-dose glucocorticoids (≤10 mg/day prednisone or equivalent) for adrenal insufficiency are allowed;
* Major surgery within 28 days prior to the first dose (excluding diagnostic surgery), or anticipated major surgery during the study (excluding diagnostic surgery); diagnostic or minimally invasive surgery within 7 days prior to the first dose;
* Live attenuated vaccines within 28 days prior to the first dose, or anticipated need for live attenuated vaccines during the study (patients are not allowed to receive live attenuated influenza vaccines within 28 days prior to the first dose, during treatment, or within 5 months after adebelimab);
* Patients with a history of allogeneic bone marrow transplantation or solid organ transplantation;
* Known allergy, hypersensitivity, or intolerance to adebelimab, other monoclonal antibodies, apatinib, chemotherapy drugs, or their excipients;
* Known psychiatric disorders, alcoholism, drug abuse, or substance abuse;
* Other factors that, in the investigator's judgment, may lead to premature termination of the study, such as non-compliance with the protocol, other severe diseases (including psychiatric disorders) requiring concomitant treatment, significant laboratory abnormalities, or family/social factors that may affect the patient's safety or data/sample collection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
PFS assessed by the investigator | From enrollment to 3 years
  PFS (Progression-Free Survival) is defined as the period of time from the start of treatment to disease progression or death from any cause.

SECONDARY OUTCOMES:
Overall Survival | From enrollment to 5 years
  OS defined as the period of time from the start of treatment to death of the patient from any cause.
AEs | From enrollment to 5 years
  Including treatment-related adverse events (AEs), serious adverse events (SAEs); the incidence of AEs and SAEs related to the study drugs (assessed according to the NCI CTCAE 5.0 criteria).
Quality of life assessed using the EORTC QLQ-C30 | From enrollment to 5 years
  The symptoms and health-related quality of life of patients will be assessed using the EORTC QLQ-C30
Quality of life assessed using the QLQ-LC13 | From enrollment to 5 years
  The symptoms and health-related quality of life of patients will be assessed using the QLQ-LC13.

OTHER OUTCOMES:
Biomarker | From enrollment to 5 years
  Exploration of potential biomarkers (PD-L1, ctDNA, CTC, NSE, etc.)

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No